CLINICAL TRIAL: NCT00786747
Title: Randomized Controlled Trial of Tailored Interactive Multimedia to Reduce Colorectal Cancer Screening Disparities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: University of Rochester (Other); City University of New York, School of Public Health (Other)
Responsible Party: Principal Investigator, Anthony F. Jerant, Professor, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: NCI -1R01CA131386-01A1; ARRA CA13138602S1 (Other Grant/Funding Number: American Reinvestment and Recovery Act supplement)
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Colorectal Neoplasms
Keywords: Computer-assisted instruction; Health knowledge, attitudes, practice; Mass screening; Patient acceptance of health care; Patient education as topic; Primary health care; Self-efficacy
MeSH Terms: conditions — Colorectal Neoplasms; Behavior; Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personally tailored computer program (Experimental): The experimental computer program provides the user with information about colorectal cancer screening that is tailored to their self-efficacy, readiness, and perceived barriers to undergoing screening, in their preferred language (English or Spanish).
  Interventions: Behavioral: Personally tailored computer program
- Non-tailored control computer program (Active Comparator): This program provides non-tailored, generic information about colorectal cancer screening, in the user's preferred language (English or Spanish).
  Interventions: Behavioral: Non-tailored control computer program

INTERVENTIONS:
Behavioral: Personally tailored computer program — The experimental computer program provides the user with information about colorectal cancer screening that is tailored to their self-efficacy, readiness, and perceived barriers to undergoing screening, in their preferred language (English or Spanish).
  Arms: Personally tailored computer program
Behavioral: Non-tailored control computer program — This program provides users with non-tailored information about colorectal cancer screening, in their preferred language (English or Spanish).
  Arms: Non-tailored control computer program

SUMMARY:
The study investigators have developed an interactive multimedia computer program that provides personally tailored education about colorectal cancer screening in the user's preferred language (English or Spanish). In this study, the investigators will examine whether use of the computer program increases the number of Hispanic patients who receive colorectal cancer screening and lessens or eliminates the glaring disparity in screening between Hispanics and non-Hispanic whites.

DETAILED DESCRIPTION:
* Background: Interactive multimedia computer programs (IMCPs) show promise as a way of delivering personally tailored (PT) information to enhance cognitive mediators of health behavior and improve patient outcomes. However, it is unclear whether PT IMCPs can be deployed in primary care offices to increase cancer screening uptake and eliminate ethnic disparities in uptake by providing PT information in each user's preferred language.
* Aims/Hypotheses: We will compare changes in colorectal cancer (CRC) screening cognitive mediators (self-efficacy, perceived barriers, and readiness) and uptake resulting from an IMCP - PT to enhance the key cognitive mediators and targeted to patients' self-identified ethnicity - with changes resulting from a non-tailored "electronic leaflet" control IMCP. The experimental and control IMCPs will each be offered in English and Spanish versions. We hypothesize that, compared with the appropriate control condition (English, Spanish, or both combined): (1) the English version of the PT IMCP will enhance the cognitive mediators of CRC screening behavior for English-speaking Hispanics and non-Hispanics; (2) there will be similarly favorable changes in these mediators for Hispanics using the Spanish version of the PT IMCP; (3) deployment of the PT IMCP will provide evidence of elimination of disparities in CRC screening between Hispanic and non-Hispanic subjects via its relative impact on the cognitive mediators in these groups; and (4) the PT IMCP (English and Spanish combined) will increase CRC screening uptake in Hispanics and non-Hispanics (considered separately) via changes in the cognitive mediators.
* Methods: Randomized controlled trial of 2 groups, comparing a PT (to the cognitive mediators) CRC screening IMCP offered in both English and Spanish versions and deployed before a primary care office visit with a non-tailored "electronic leaflet" CRC screening IMCP (control) also offered in both English and Spanish. Screening methods targeted will be fecal occult blood testing, flexible sigmoidoscopy, and colonoscopy. Primary outcomes will be CRC screening uptake, self-efficacy, perceived barriers, and readiness.
* Implications: Our findings will determine whether an IMCP that is PT to cognitive mediators of screening behavior and deployed in primary care offices prior to previously scheduled visits can activate patients of various ethnicities to undergo CRC screening. They may also suggest a promising, portable method of reducing disparities in CRC (and other) screening uptake between Hispanic and non-Hispanic individuals.

ELIGIBILITY:
Inclusion Criteria:

* Receive primary care at one of the participating outpatient study offices
* Age at or above 50 years
* Able to read and speak English and/or Spanish
* Adequate vision, hearing, and hand function to use an IMCP running on a laptop computer via a touch screen interface
* Have an active telephone
* Not up to date for CRC screening. Up to date status will be defined as having completed CRC screening via: fecal occult blood test within 2 years; flexible sigmoidoscopy within 5 years; or colonoscopy within 10 years, consistent with national practice guidelines and standards.

Exclusion Criteria:

* Unable to understand the consent form or the telephone screening questionnaire due to cognitive impairment
* Unable to provide informed consent due to serious acute illness

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1164 (Actual)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Up to date colorectal cancer screening status | 1 year

SECONDARY OUTCOMES:
Up to date colonoscopy screening status | 1 year
Up to date fecal occult blood testing status | 1 year
Colorectal cancer screening self-efficacy | Immediately after computer program use
Perceived barriers to colorectal cancer screening | Immediately after computer program use
Readiness to undergo colorectal cancer screening | Immediately after computer program use

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Jerant, MD, Principal Investigator — University of California, Davis
Locations (5):
- United States (5):
  - University of California, Davis Health System, Sacramento, California
  - University of Colorado, Aurora, Colorado
  - Sophie Davis School of Biomedical Education, City University of New York,, New York, New York
  - University of Rochester School of Medicine and Dentistry, Rochester, New York
  - University of Texas Health Sciences Center, San Antonio, Texas

REFERENCES:
- [Background] Sohler NL, Jerant A, Franks P. Socio-psychological factors in the Expanded Health Belief Model and subsequent colorectal cancer screening. Patient Educ Couns. 2015 Jul;98(7):901-7. doi: 10.1016/j.pec.2015.03.023. Epub 2015 Apr 8. PMID 25892503
- [Background] Jerant A, Sohler N, Fiscella K, Franks B, Franks P. Tailored interactive multimedia computer programs to reduce health disparities: opportunities and challenges. Patient Educ Couns. 2011 Nov;85(2):323-30. doi: 10.1016/j.pec.2010.11.012. Epub 2010 Dec 13. PMID 21146950
- [Result] Jerant A, Kravitz RL, Sohler N, Fiscella K, Romero RL, Parnes B, Tancredi DJ, Aguilar-Gaxiola S, Slee C, Dvorak S, Turner C, Hudnut A, Prieto F, Franks P. Sociopsychological tailoring to address colorectal cancer screening disparities: a randomized controlled trial. Ann Fam Med. 2014 May-Jun;12(3):204-14. doi: 10.1370/afm.1623. PMID 24821891
- [Result] Jerant A, Kravitz RL, Fiscella K, Sohler N, Romero RL, Parnes B, Aguilar-Gaxiola S, Turner C, Dvorak S, Franks P. Effects of tailored knowledge enhancement on colorectal cancer screening preference across ethnic and language groups. Patient Educ Couns. 2013 Jan;90(1):103-10. doi: 10.1016/j.pec.2012.08.017. Epub 2012 Sep 15. PMID 22985627
- [Result] Jerant A, To P, Franks P. The effects of tailoring knowledge acquisition on colorectal cancer screening self-efficacy. J Health Commun. 2015;20(6):697-709. doi: 10.1080/10810730.2015.1018562. Epub 2015 Apr 30. PMID 25928315